CLINICAL TRIAL: NCT05323955
Title: Secondary BRain Metastases Prevention After Isolated Intracranial Progression on Trastuzumab/Pertuzumab or T-DM1 in Patients With aDvanced Human Epidermal Growth Factor Receptor 2+ brEast Cancer With the Addition of Tucatinib
Acronym: BRIDGET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carey Anders, M.D. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Carey Anders, M.D., Sponsor Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109777
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Brain Metastases; Human Epidermal Growth Factor 2 Positive Carcinoma of Breast; Advanced Breast Cancer
Keywords: Brain metastases; HER2+ breast cancer; Trastuzumab; Pertuzumab; T-DM1
MeSH Terms: conditions — Brain Neoplasms | interventions — Trastuzumab; Ado-Trastuzumab Emtansine; pertuzumab; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Trastuzumab/pertuzumab + tucatinib or T-DM1 + tucatinib
  300mg of tucatinib taken orally twice a day. Taken on Days 1-21 of a 21 Day cycle (3 Weeks).
  Trastuzumab/Biosimilar administered per current package insert based on site standard of care guidelines
  Pertuzumab or Biosimilar administered per current package insert based on site standard of care guidelines
  Trastuzumab Emtansine (T-DM1) administered per current package insert based on site standard of care guidelines
  Interventions: Drug: Trastuzumab; Drug: Trastuzumab Emtansine (T-DM1); Drug: Pertuzumab; Drug: Tucatinib

INTERVENTIONS:
Drug: Trastuzumab — Administer per current package insert based on site standard of care guidelines
  Other Names: Herceptin
Drug: Trastuzumab Emtansine (T-DM1) — Administer per current package insert based on site standard of care guidelines
Drug: Pertuzumab — Administer per current package insert based on site standard of care guidelines
  Other Names: Perjeta
Drug: Tucatinib — 300 mg orally twice daily (21 Day Cycle)
  Other Names: Tukysa

SUMMARY:
Patients with advanced HER2+ breast cancer on maintenance trastuzumab/pertuzumab or T-DM1 with 1st or 2nd intracranial disease event (brain metastases) and stable extracranial disease will be enrolled. They will receive local therapy with stereotactic radiosurgery ± surgical resection if indicated followed by enrollment. Patients will continue standard of care trastuzumab/pertuzumab or T-DM1 with the addition of tucatinib. Hormone receptor positive patients requiring endocrine therapy should continue. Study treatment will continue until disease progression or intolerable side effects. Patients on trial with extracranial disease progression with stable intracranial disease should continue tucatinib into next line of therapy.

DETAILED DESCRIPTION:
Patients with advanced HER2+ breast cancer on either (1) first-line trastuzumab/pertuzumab OR (2) second-line T-DM1 in the metastatic setting OR (3) adjuvant trastuzumab-based therapy or T-DM1 with isolated intracranial recurrence will be included. Patients with de novo metastatic disease and brain metastases or isolated intracranial recurrence can enter upon initiation of maintenance trastuzumab/pertuzumab after chemotherapy if deemed necessary by treating oncologist and meeting other inclusion criteria. Patients with 1st or 2nd intracranial disease event (brain metastases) and stable extracranial disease will be enrolled. Third intracranial progression would be considered if > 12 month interval between second and third intracranial progression. They will receive local therapy with stereotactic radiosurgery ± surgical resection followed by enrollment. Patients will continue standard of care treatment trastuzumab/pertuzumab or T-DM1 with the addition of tucatinib. Hormone receptor-positive patients requiring endocrine therapy should continue.

Study treatment will continue until intercranial disease progression or intolerable side effects. Patients with extracranial disease progression while on trial with stable intracranial disease should continue tucatinib into the next line of therapy as described in protocol. If a subject continues tucatinib into the next line therapy they are still considered on study treatment and will be monitored according to the protocol. Cycles will continue consecutively and not restart. Once the subject comes off tucatinib they are considered off study treatment and will enter the follow up period.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Locally advanced/unresectable or metastatic breast cancer with presence of brain metastases (Stage IV).
* Histologically confirmed HER2+ breast carcinoma by ASCO-CAP guidelines, with HER2+ defined by in situ hybridization (ISH), immunohistochemistry (IHC), or fluorescence in situ hybridization (FISH) methodology on most recent biopsy (primary tissue).
* Currently receiving: (1) first-line trastuzumab/pertuzumab with or without endocrine therapy OR (2) second-line T-DM1 in the metastatic setting OR (3) adjuvant trastuzumab-based therapy or T-DM1 with isolated intracranial recurrence. Patients with de novo metastatic disease and brain metastases or isolated metastatic disease to the brain can enroll at time of initiation of trastuzumab/pertuzumab. Induction taxane therapy is not required and need to administer can be determined by the treating physician. Patients on trastuzumab alone are allowed if pertuzumab not tolerated.
* Systemic disease otherwise stable per RECIST 1.1 or no evidence of extracranial disease.
* Adequate hepatic and renal function and hematologic parameters:

  * Absolute neutrophil count (ANC) ≥ 1.0 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 9 g/dL
  * Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases are present)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min as calculated using the Cockcroft-Gault (CG) equation
  * Left ventricular ejection fraction (LVEF) ≥ 50%.
* Central nervous system inclusion - Based on screening brain magnetic resonance imaging (MRI), patients must have ALL of the following:

  * Adequate local therapy to existing brain lesions ≥ 5mm including surgical resection and/or stereotactic radiosurgery
  * Limited to first or second intracranial progression. Third intracranial progression would be considered if > 12 month interval between second and third intracranial progression.
  * Time since stereotactic radiosurgery (SRS) is ≥ 7 days prior to first dose of study treatment.
  * Time since surgical resection is ≥ 14 days prior to first dose of study treatment.
  * Time since local therapy < 12 weeks. Patients with de novo metastastic breast cancer presenting with brain metastases may enter following cessation of chemotherapy if within 24 weeks of local therapy to the brain and brain metastases have remained stable based on brain MRI.
  * Prior radiation is required within 12 weeks of enrollment to at least 1 brain lesion. Other brain lesions under 5mm do not require treatment.

NOTE: Relevant records of any CNS treatment including radiation must be available to allow for classification of target and non-target lesions

* Females of childbearing potential must have a negative serum pregnancy test at screening. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential and males must be willing to abstain from heterosexual intercourse or to use contraception as outlined in the protocol.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Previously been treated with: Lapatinib, neratinib, afatinib, tucatinib or other investigational HER2/epidermal growth factor receptor (EGFR) or HER2 tyrosine kinase inhibitor (TKI) at any time previously (patients treated with adjuvant neratinib allowed if relapse > 12 months after last dose).
* Clinically significant cardiopulmonary disease.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including:

  * tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice),
  * hepatitis B (known positive HBV surface antigen (HBsAg) result),
  * hepatitis C, or
  * human immunodeficiency virus (positive HIV 1/2 antibodies)

NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed if they are stable and have been on treatment for ≥ 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required.

* Unable for any reason to undergo MRI of the brain
* Use of a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor, or a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment. See protocol.
* Central nervous system exclusion - Based on screening brain MRI, patients must not have any of the following:

  * Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent)
  * Diffuse leptomeningeal disease or positive CSF cytology; however, discreet dural-based metastases are allowed
  * Poorly controlled seizures. Defined as seizures that continue to occur despite optimal anticonvulsant medications based on investigator discretion.
  * History of whole brain radiation therapy
  * Any untreated brain lesions ≥ 5 mm
* Active infection requiring intravenous systemic therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Patients with a prior or concurrent malignancy within last 3 years whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.
* Treatment with any investigational drug within 30 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 3 years
  Evaluate the ability of tucatinib in combination with trastuzumab/pertuzumab or TDM-1 to prolong intracranial progression free survival (PFS) in patients compared to historical controls. PFS is defined as the time from the day of study treatment initiation until evidence of intracranial disease progression per RANO-BM or death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival by RECIST 1.1 | 3 years
  Evaluate the progression free survival by RECIST 1.1 criteria. PFS is defined as time from the day of study treatment initiation until evidence of disease progression per RECIST v1.1 or death from any cause.
Progression Free Survival of Extracranial Disease | 3 years
  Evaluate PFS of extracranial disease. PFS is defined as time from the day of study treatment initiation until evidence of extracranial disease progression per RECIST v1.1 or death from any cause.
Distant Versus Local Intracranial Progression Free Survival | 3 years
  Evaluate distant versus local intracranial PFS.
Site of First Progression | 3 years
  Evaluate the site of first progression (CNS vs non-CNS). Site of first progression (CNS vs non-CNS) is defined by first site of progression on trial either within the central nervous system or extracranial disease as defined by investigator
Overall Survival (OS) | 3 years
  Evaluate OS. OS defined as day of study treatment initiation until death from any cause.
Assess Adverse Events | 2 months
  Evaluate the toxicity profile of agents in patients with brain metastases. Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Carey Anders, MD, Principal Investigator — Duke Cancer Institute
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No